CLINICAL TRIAL: NCT06180031
Title: Effect of Adding Magnesium Sulphate to Bupivacaine in Ultrasound Guided Pericapsular Nerve Group Block for Post Operative Analgesia in Hip Joints Surgeries
Brief Title: Effect of Adding Magnesium Sulphate in Pericapsular Nerve Group Block
Acronym: Peng Block
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mustafa Mahmoud Muhammed Bekhet, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04-2023-200535
Record Dates: First submitted 2023-12-02; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (control) (No Intervention): will have Peng block using 20mg bupivacaine 0.25%
- Group M (Active Comparator): will have PENG block with 2mg magnesium sulphate 10% as an adjuvant to 20mg of bupivacaine 0.25%
  Interventions: Drug: Pericapsular nerve group block using bupivicaine and magnesium sulphate

INTERVENTIONS:
Drug: Pericapsular nerve group block using bupivicaine and magnesium sulphate — This technique involves the deposition of the local anesthetic in the fascial plane between the psoas muscle and the superior pubic ramus
  Arms: Group M

SUMMARY:
Our aim will be to compare the analgesic efficacy and safety of magnesium sulphate as an adjuvant to bupivacaine in pericapsular nerve group block in Hip joint surgeries.

* Our primary outcome of the study: total amount of postoperative morphine consumption in the first 24h postoperative.
* Our secondary outcome of the study: mean arterial blood pressure, heart rate, respiratory rate, adverse effects, block related complication, sedation score (by Ramsay sedation scale) and pain score (by Visual Analog Scale)

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged 18 years or more.

  * Patients with American society of anesthesiologists (ASA) classification class I or II
  * Patients weight range from 50 to 90 Kgs

Exclusion Criteria:

* • Patient refusal of peripheral nerve block

  * Patient with infection at the site of injection
  * Patient with coagulopathy
  * Patients with known allergy to used medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain management | 24 hours postoperatively
  total amount of postoperative morphine consumption in the first 24 hours postoperatively.

SECONDARY OUTCOMES:
Visual analog scale | 24 hours postoperatively
  It's a scale from 0 to 10 where 0 means no pain and 10 means worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Attia, Professor, Study Chair — Assiut University; Fatma A Abd Diab, Associate Professor, Study Director — South Egypt's cancer institute, Assiut University; Moaz Tohamy, Lecturer, Study Director — South Egypt's cancer institute, Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt